CLINICAL TRIAL: NCT06047938
Title: Familial Mediteranean Fever in Upper Egypt, and Its Relation to Atherosclerosis in Children
Brief Title: FMF and Atheroscelerosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali AbdElhaleem Hussein, Doctor, Assiut University
Other Study IDs: FMF and atheroscelerosis
Record Dates: First submitted 2023-07-12; First posted 2023-09-21 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: FMF

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- carotid intima thickness measurment: CIT will be assessed using ultrasound evaluation by measuring the intima-media thickness of carotid arteries (IMT). This non-invasive method is used to detect subclinical atherosclerosis and it can be used in a multitude of patients including children. It will be carried out on the two study groups (FMF patients and the control group) and the results will be compared. It will be conducted in Assiut University Neurosonology Unit, at the Department of Neurology.
  Interventions: Radiation: ultrasound on carotid

INTERVENTIONS:
Radiation: ultrasound on carotid — CIT will be assessed using ultrasound evaluation by measuring the intima-media thickness of carotid arteries (IMT). This non-invasive method is used to detect subclinical atherosclerosis and it can be used in a multitude of patients including children[11]. It will be carried out on the two study groups (FMF patients and the control group) and the results will be compared. It will be conducted in Assiut University Neurosonology Unit, at the Department of Neurology.

SUMMARY:
The aim of this study is to search for subclinical atherosclerosis in children diagnosed as FMF in Assiut University children's Hospital, and to correlate the risk to develop atherosclerosis to the different characters and genetic variants of FMF.

DETAILED DESCRIPTION:
* To describe the clinical characteristics of patients diagnosed as FMF in Upper Egypt, and to find the most common presenting symptoms.
* To mention the most common genetic variants reported in FMF patients in Upper Egypt, and to correlate the genetic variant with the risk to develop atherosclerosis.
* To assess the growth parameters in patients with FMF and compare it with the control group.
* To estimate the differences in Complete blood count (CBC) parameters, lipid profile, CIT in patients with FMF and control group.
* To search for subclinical atherosclerosis in patients with FMF based on their lipid profile and CIT.

ELIGIBILITY:
Inclusion Criteria:

1. Age at enrollment less than18 years.
2. Both sexes.
3. Diagnosed as familial Mediterranean fever according to Tel Hashomer criteria. [10]

Exclusion Criteria:

1. Patients with acute or chronic active infections.
2. Patients with pre-existing illness as chronic lung, liver or renal diseases.
3. Patients with diabetes mellitus, atherosclerotic vascular disease.
4. Patients with malignancy

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All patients that present with FMF in Assiut University Pediatric Hospital (allergy , immunology and rheumatology department)in one year.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2024-09-14 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
detecting subclinical atheroscelerosis | It will be measured in one year
  The aim of this study is to detect subclinical
  atherosclerosis in children diagnosed as FMF in Assiut University children's Hospital by measuring carotid intima thickness